CLINICAL TRIAL: NCT00904657
Title: An Open-label One-way Explorative Study on the Pharmacokinetics and Pharmacodynamics of Sunitinib in Healthy Volunteers
Brief Title: An Explorative Study on the Pharmacokinetics and Pharmacodynamics of Sunitinib in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: University Hospital, Bonn (Other); ZKS Köln (Other)
Responsible Party: Prof. Dr. Med. U. Fuhr, University of Cologne
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Uni-Koeln-1127
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2009-12

CONDITIONS: Blood Pressure
Keywords: pharmacokinetic/pharmacodynamic modeling; biomarkers (growth factors) as a possible tool of drug effect
MeSH Terms: interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: sunitinib (Sutent) — 50 mg capsule Sutent, one application a day for five days

SUMMARY:
The study is conducted:

* to investigate the influence of sunitinib (study drug) on the plasma biomarkers VEGF-A, VEGF-C, soluble VEGFR-2, and soluble VEGFR-3 (vessel endothelial growth factors) and on the blood pressure;
* to generate a pharmacokinetic/pharmacodynamic model for sunitinib using biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* Male/Female
* Age: 18-55 years
* Body weight of 60 kg or higher, Body Mass Index 19 - 27 kg/m2
* Considered to be healthy on the basis of extensive pre-study screening
* Willing and capable to confirm written consent to enrolment after ample information has been provided

Exclusion Criteria:

* Ongoing healing of wound or parenchymal tissue requiring angiogenesis
* Any skin abnormality and/or neurodermatitis and /or chronic skin disease
* A history of haemorrhage
* A history of any gastrointestinal event with persisting clinical relevance
* A history of pancreatitis
* History of cerebrovascular accident or transient ischemic attack or seizures
* History of pulmonary embolism
* History of venous thromboembolic events
* History of hypertension
* A history of cardiac events within 12 months prior to sunitinib administration such as myocardial infarction (including severe/unstable angina), coronary/peripheral artery bypass graft
* Any relevant clinical abnormality (as based on extensive medical history, amination, vital signs and 12-lead ECG)
* Inadequate cardiac function [left ventricular ejection fraction (LVEF) < lower limit of normal (LLN) as assessed by echocardiography (ECHO)]
* A history of any surgical abdominal intervention (including appendectomy) or of peritonitis
* Bronchial asthma, COPD, or actual obstructive bronchitis
* Hypothyroidism /hyperthyroidism
* Cardiac insufficiency
* Liver disease
* Cardiac dysrhythmia (e.g., prolongation of the QT interval)
* Diabetes mellitus
* Chronic infections
* Relevant acute infections or with actual therapy-requiring allergies (including drug allergies) within the last two weeks
* Suspicion of hypersensitivity to sunitinib or to any of the excipients
* Any clinically relevant laboratory abnormality
* Subjects receiving any medication within 2 weeks prior to study start or during the study (exceptions possible upon decision of Principal Investigator, e.g., paracetamol (acetaminophen) single dose for acute pain or topical aciclovir for herpes simplex)
* Subjects who have taken a drug with a long half-life (> 24 hours) within four weeks before the first trial day
* Subjects who received chronic drug treatment (> 3 days) within eight weeks before the first trial day
* Subjects who participated in a clinical trial within the last 3 months before the start of the present study
* Subjects who donated blood or plasma within the last 12 weeks before the start of the present study
* Subjects who smoke, i.e., subjects who smoked one or more cigarettes during the last six months
* Subjects who are known or suspected to be (social) drug dependent, incl. those drinking more than 30 g alcohol per day
* Subjects with a history of alcohol or recreational drug addiction
* Subjects with a history of any severe disease that might interfere with the study objectives (e.g. psychiatric disease, epilepsy)
* Subjects who are not willing or able to abstain from alcohol, methylxanthine-containing beverages and foods, and grapefruit flesh/juice for 72 hours before first study drug administration until 2 weeks after last study drug administration
* Subjects who adhere to a special diet (e.g., vegetarians) or lifestyle (including working at night and extreme physical activities such as competitive sports and weight lifting) that might interfere with the investigation
* Subjects planning elective hospital treatment within two months after last intake of trial medication
* Subjects who are known or suspected not to comply with the study directives and/or known or suspected not to be reliable or trustworthy
* Subjects who are known or suspected not to be capable of understanding and evaluating the information that is given to them as part of the formal information policy (informed consent), in particular regarding the foreseeable risks and discomfort to which they will be exposed
* Subjects with anticipated problems of successfully placing an indwelling venous catheter at a forearm
* Female subjects only:

  * positive results in pregnancy test
  * pregnant and lactating women
  * subjects who do not use or does not agree to use appropriate contraceptive methods during the study and two months after the study
* Male subjects only: they have to accept not to procreate children during the study and two months after the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)